CLINICAL TRIAL: NCT01821261
Title: Three Month Clinical Efficacy of an Ethyl Lauroyl Arginate HCL (LAE) Mouth Rinse: Effect on Gingivitis
Brief Title: A Clinical Trial to Test the Effect of an Experimental Mouth Rinse on Gum Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LAEBBA0004
Record Dates: First submitted 2013-03-22; First posted 2013-03-29 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Gingivitis
Keywords: Gums; Gingiva; Gingival Inflammation; Gingival Bleeding
MeSH Terms: conditions — Gingivitis; Gingival Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Mouth Rinse 19668-012 (Experimental): Twice each day, brush with about one inch of toothpaste 035000513007 in the usual manner, rinse mouth with water, and then rinse with 20 ml of mouth rinse 19668-012 for 30 seconds and spit it out - do not swallow.
  Interventions: Device: Mouth Rinse 19668-012; Drug: Toothpaste 035000513007
- Mouth Rinse 500347078842 (Active Comparator): Twice each day, brush with about one inch of toothpaste 035000513007 in the usual manner, rinse mouth with water, and then rinse with 10 ml of mouth rinse 500347078842 for 60 seconds and spit it out - do not swallow.
  Attention: Toothpastes can stop mouth rinse from working. Rinse your mouth thoroughly with water and wait 5 minutes after brushing your teeth before using the mouth rinse. You can also use the mouthwash at a different time of day.
  Interventions: Drug: Mouth Rinse 500347078842; Drug: Toothpaste 035000513007
- Toothpaste 035000513007 (Other): Twice each day, brush with about one inch of toothpaste 035000513007 in the usual manner. Subjects in this arm will not use any mouth rinse.
  Interventions: Drug: Toothpaste 035000513007

INTERVENTIONS:
Device: Mouth Rinse 19668-012 — 20 ml of experimental mouth rinse 19668-012 for 30 seconds, twice daily
  Arms: Mouth Rinse 19668-012
Drug: Mouth Rinse 500347078842 — 10 ml of mouth rinse 500347078842 for 60 seconds, twice daily
  Other Names: Mouth rinse containing Chlorhexidine; Corsodyl Mouthwash
  Arms: Mouth Rinse 500347078842
Drug: Toothpaste 035000513007 — Approximately one inch of toothpaste 035000513007, twice daily
  Other Names: Toothpaste containing fluoride; Colgate® Cavity Protection Regular

SUMMARY:
Subjects will be given special instructions about eating, smoking and taking care of their teeth during the 18 hours before they come to the dentist's office for screening. At that first visit, they will be examined by a dentist, who will examine their mouths with a dental instrument to determine whether they qualify to participate in the trial. Someone who works for the dentist will also take some oral measurements.

Participants who qualify to be in the study will receive a treatment for their gingivitis and have an equal chance of being assigned to one of three treatment groups. Subjects in all three groups will be given toothpaste that is already available in stores. They will brush their teeth twice daily with a one-inch strip of toothpaste in their regular manner. After brushing, subjects in one group will use an experimental mouth rinse that is not available in stores. Another group will be given a mouth rinse to use that is already available in stores, and the third group will not use any mouth rinse at all. After they receive their assigned products subjects will be supervised while they brush their teeth and/or rinse to ensure they understand exactly how to use the products. All other brushing and rinsing over the next three months will be at home, but subjects will be required to keep a diary to record their brushing and rinsing times twice each day.

Subjects will be required to bring their diaries and any leftover toothpaste and mouth rinse with them for four more scheduled appointments after about 1 week, 2 weeks, 4 weeks, and 3 months. At those appointments, the dentist will examine their mouths, make sure there are no safety concerns, and examine again to get the measurements needed. One of the dentist's staff members will take other measurements as well.

The study will determine the measured effects of the experimental mouth rinse on gingivitis, and compare these results to the mouth rinse that is already available, as well as to using no mouth rinse at all.

DETAILED DESCRIPTION:
At screening/baseline, subjects will present to the clinical site having refrained from oral hygiene for at least 8 hours, but no more than 18 hours, and from eating or smoking for at least 4 hours for baseline examinations. Baseline examinations will include Macpherson modification of the Lobene Stain Index (Extrinsic Stain), Volpe-Manhold Index (Calculus), and oral hard and soft tissue exam, Modified Gingival Index (MGI), Bleeding Index (BI) and Plaque Index (PI). After the baseline oral examinations, subjects who qualify will receive a whole-mouth supragingival dental prophylaxis and random assignment to one of three treatment groups.

Subjects randomized to the control group will brush twice daily with a marketed fluoride toothpaste. Subjects randomized to the experimental group will brush twice daily with a marketed fluoride toothpaste and use an experimental mouth rinse. The last randomized group will brush twice daily with a marketed fluoride toothpaste and rinse with a marketed mouth rinse twice daily. The first product use will be conducted under supervision of study personnel. All other brushing and rinsing will be unsupervised and the subjects will be required to maintain a diary card to document twice-daily product use, with brushing and rinsing times. Diaries along with product accountability will be used to check for subject compliance.

Subjects will return to the clinical site after one week (Day 7±1 day), two weeks (Day 14±2 days), four weeks (Day 28±3 days) and three months (Day 91±5 days). Oral hard and soft tissue safety, MGI, BI, and PI will be assessed at all visits. Extrinsic Stain and Calculus will be assessed at baseline, four weeks and three months by a different examiner.

At the end of the study, subjects will return all used and unused product to the clinical site.

ELIGIBILITY:
Inclusion Criteria:

* Assessed by site personnel as able to comprehend and follow the requirements of the study in the Portuguese language, and to be available on scheduled visit dates
* After being informed of all pertinent aspects of the trial, and having all questions answered, voluntarily signed an informed consent document
* Assessed by the investigator to have gingivitis, and otherwise qualify to be a participant in the trial

Exclusion Criteria:

* Relative, partner or staff of any clinical research site personnel
* Any oral, psychiatric or medical condition (including pregnancy or nursing), laboratory abnormality, or use of experimental or other products that may (per protocol or in the opinion of the investigator) compromise the safety of the participant or the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2014-04-30 (Estimated); Study Completion 2014-07-31 (Estimated)

PRIMARY OUTCOMES:
Whole-mouth Mean Bleeding Index (BI) at 3 Months | 3 months
  Bleeding after periodontal probe will be assessed by scores on a scale of 0-2 using the Gingival Bleeding Index (BI), where 0=Absence of Bleeding after 30 Seconds and 2=Immediate Bleeding.

SECONDARY OUTCOMES:
Whole-mouth Mean Bleeding Index (BI) | within 4 weeks
  Bleeding after periodontal probe will be assessed by scores on a scale of 0-2 using the Gingival Bleeding Index (BI), where 0=Absence of Bleeding after 30 Seconds and 2=Immediate Bleeding.
Whole-mouth Mean Modified Gingival Index (MGI) | within 3 months
  Gingivitis will be assessed by scoring inflammation on a 0-4 scale, according to the Modified Gingival Index, where 0=Normal and 4=Severe Inflammation.
Whole Mouth Mean Plaque Index (PI) | within 3 months
  Plaque will be assessed on a scale of 0-5 using the Turesky modification of the Quigley-Hein Plaque Index, where 0=No plaque and 5=Plaque covering 2/3 or more of surface.
Mean Area Stain Score for Mesial Region | within 3 months
  A mean area stain score for the Mesial Region will be recorded on a scale of 0-3, where 0 = no stain present, natural tooth color and 3 = stain outside pits/grooves, over 10% of surface affected
Mean Area Stain Score for Gingival Region | within 3 months
  A mean area stain score will be recorded for Gingival Region, on a scale of 0-3, where 0 = no stain present, natural tooth color and 3 = stain outside pits/grooves, over 10% of surface affected
Mean Area Stain Score for Distal Region | within 3 months
  A mean area stain score will be recorded for Distal Region, on a scale of 0-3, where 0 = no stain present, natural tooth color and 3 = stain outside pits/grooves, over 10% of surface affected
Mean Area Stain Score for Body of Tooth | within 3 months
  Mean area stain scores will be recorded for Body of Tooth, on a scale of 0-3, where 0 = no stain present, natural tooth color and 3 = stain outside pits/grooves, over 10% of surface affected
Mean Stain Intensity Score | within 3 months
  A score for stain intensity will be recorded on a scale of 0-3, where 0 = no stain and 3 = heavy, dark stain (obvious and aesthetically unacceptable)
Mean Tartar Height | within 3 months
  Mean tartar height will be recorded in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lynch, DMD, PhD, Study Director — Johnson & Johnson Consumer Inc. (J&JCI)